CLINICAL TRIAL: NCT03680365
Title: Your Voice; Impact of DMD. A Qualitative Assessment of the Impact of DMD on the Lives of Families
Brief Title: Your Voice; Impact of Duchenne Muscular Dystrophy (DMD) on the Lives of Families
Status: Completed | Type: Observational
Sponsor: Jett Foundation, Inc. (Other)
Collaborators: Engage Health Inc. (Industry); Hyman, Phelps, & McNamara, P.C. (Unknown); Ryans Quest Inc. (Unknown); Michaels Cause Inc. (Unknown); Nationwide Children's Hospital (Other); Solid Biosciences Inc. (Industry); Santhera Pharmaceuticals (Industry); Italfarmaco (Industry); Catabasis Pharmaceuticals (Industry); Wave Life Sciences Ltd. (Industry); Sarepta Therapeutics, Inc. (Industry); Hoffmann-La Roche (Industry); Pfizer (Industry); Capricor Inc. (Industry); NS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Jett 0001
Record Dates: First submitted 2018-09-06; First posted 2018-09-21 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Duchenne Muscular Dystrophy; Burden, Dependency; Disability Physical; Disease Management; Impairment; Rare Diseases
Keywords: Duchenne, DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to improve the understanding of the treatment goals that a person with Duchenne Muscular Dystrophy (DMD) or the caregiver may be most interested in, based on the severity of the person's disease. Data will be collected by online survey when the participant accepts the study invitation ("RSVP questionnaire") and telephone interview on the functional burden and self-identified treatment goals from the perspective of people with DMD and their caregivers. Interviews will be analyzed to help identify things important to Duchenne families to measure in clinical trials and to inform the selection of key concepts of interest and development of future clinical outcome measures, including observer reported outcomes/patient reported outcomes. The study will be conducted in the United States and will enroll between 45 and 120 participants 11 years or older living with DMD as well as their caregivers. The time commitment for the online survey and the telephone interview is about one hour. It is anticipated that the entire study will be completed within one year.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a person with DMD who is 11 years or older or The parent/legal guardian of a person with DMD who is under the age of 18 years.
2. Confirmed diagnosis of DMD with written proof of disease provided
3. Resident of the U.S.
4. Able to read, write and communicate in English
5. Able to grant informed consent
6. Willing to participate in a 45 minute telephone interview
7. Ability to view or receive a document from the interviewer before or during the interview (web browser, ability to receive a text, fax or document by mail)

Exclusion Criteria:

1. Inability to meet any of the inclusion criteria

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in individuals 11 years or older living with Duchenne Muscular Dystrophy as well caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Patient/Parent Interview Assessing Treatment Needs | 1 year
  In this non-interventional study, up to 120 patients/parents will participate in an online survey designed to determine the patient's functional category; ambulatory, transitional, or non-ambulatory. 15 patients from each functional category will be interviewed to gather qualitative input, in the patient's voice, regarding activities they would like to do but cannot do because of DMD, and reasons why these activities are important to them. Qualitative responses will be scored to provide quantitative frequency counts and point values for each answer dependent upon if the response was the most important, 2nd most important and 3rd most important activity to the participant. Data will be coded by two independent coders to ensure consistency. Scores will be calculated by functional category for:
  1. Number of times each activity is mentioned
  2. Overall score for each activity
  3. Number of times each reason is mentioned
  4. Overall score for each reason

CONTACTS AND LOCATIONS:
Overall Officials: Christine McSherry, R.N., Principal Investigator — Jett Foundation, Inc.
Locations (1):
- Engage Health, Inc., Eagan, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989
- [Background] Birnkrant DJ, Bushby K, Bann CM, Alman BA, Apkon SD, Blackwell A, Case LE, Cripe L, Hadjiyannakis S, Olson AK, Sheehan DW, Bolen J, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: respiratory, cardiac, bone health, and orthopaedic management. Lancet Neurol. 2018 Apr;17(4):347-361. doi: 10.1016/S1474-4422(18)30025-5. Epub 2018 Feb 3. PMID 29395990
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Colvin MK, Cripe L, Herron AR, Kennedy A, Kinnett K, Naprawa J, Noritz G, Poysky J, Street N, Trout CJ, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 3: primary care, emergency management, psychosocial care, and transitions of care across the lifespan. Lancet Neurol. 2018 May;17(5):445-455. doi: 10.1016/S1474-4422(18)30026-7. Epub 2018 Feb 2. PMID 29398641
- See also: Jett Foundation — https://www.jettfoundation.org/